CLINICAL TRIAL: NCT04365218
Title: A Phase I Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of MEDI8367 Administered as Single Ascending Doses in Healthy Subjects, and as a Single Dose in Healthy Subjects of Japanese-descent and in Subjects With Chronic Kidney Disease
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics With MEDI8367 Administered in Healthy Subjects, and in Subjects With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D6361C00001
Record Dates: First submitted 2020-03-30; First posted 2020-04-28 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease
Keywords: First-in-human, Single Ascending Dose
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is blinded for subjects, Investigator and site staff, and Contract Research Organization staff with regard to treatment (MEDI8367 or placebo) at each dose level. The Sponsor will be unblinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Dose A) (Experimental): 6 subjects will be randomized to receive MEDI8367 Dose A and 2 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo
- Cohort 2 (Dose B) (Experimental): 6 subjects will be randomized to receive MEDI8367 Dose B and 2 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo
- Cohort 3 (Dose C) (Experimental): 6 subjects will be randomized to receive MEDI8367 Dose C and 2 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo
- Cohort 4 (Dose D) (Experimental): 6 subjects will be randomized to receive MEDI8367 Dose D and 2 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo
- Cohort 5 (Dose D) (Experimental): 6 subjects will be randomized to receive MEDI8367 Dose D or the highest tolerable dose based on Cohorts 1 to 4 and 2 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo
- Cohort 6 (Dose D) (Experimental): 15 subjects will be randomized to receive MEDI8367 Dose D or the highest tolerable dose based on Cohorts 1 to 4 and 15 subjects will be randomized to receive placebo.
  Interventions: Drug: MEDI8367; Drug: Placebo

INTERVENTIONS:
Drug: MEDI8367 — Subjects will receive subcutaneous (SC) single dose of MEDI8367, depending upon dose escalation strategy and Safety Review Committee results. The maximum dose will not exceed 600 mg. The dose will be administered as a single injection or multiple injections in the abdomen region.
Drug: Placebo — Saline solution for injection and the placebo volume to be administered will be equivalent to the MEDI8367 volume administered for each dosing cohort.

SUMMARY:
This Phase I First in Human (FIH) study is being conducted to determine the safety, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity profile of MEDI8367 across the dose range.

DETAILED DESCRIPTION:
This is a Phase I, FIH, randomized, blinded, placebo-controlled study, to evaluate the safety and PK of MEDI8367 as single ascending doses (SAD) in healthy subjects and as a single dose in healthy subjects of Japanese-descent and in subjects with chronic kidney disease (CKD).

Six cohorts, Cohorts 1 to 5 (healthy volunteers including Japanese subjects in Cohort 5) each consisting of 8 subjects (total 40 subjects), and Cohort 6 (subjects with CKD) consisting of 30 subjects, will participate in the study. The starting dose is dose A of MEDI8367 with up to 3 dose escalations planned (provisional doses of dose B, dose C, and dose D).

The study will comprise of:

* A Screening Period of maximum 28 days;
* A Treatment Period during which subjects will be resident at the Clinical Unit/non-clinical sites from the day before investigational medicinal product (IMP) administration (Day -1) until at least 72 hours after IMP administration; discharged on Day 4; and
* A Follow-up Period (out-patient) with 8 visits; the final Follow-up Visit (Visit 10) within 90 ± 4 days after the last IMP dose. The study day for the last visit may be adjusted based on PK/PD results from the current and previous cohorts.

Dosing for Cohorts 1 to 4 and Cohort 6 will proceed with 2 subjects in a sentinel cohort, such that one subject will be randomized to receive MEDI8367 and one subject will be randomized to receive placebo. The blinded safety data from the sentinel subjects up to 3 days post-dose will be reviewed by the site Principal Investigator (PI) before the remaining subjects in the cohort are dosed. Dosing is proposed to continue based on a lack of significant safety findings in the first 2 subjects dosed per cohort. The remaining 6 subjects in Cohorts 1 to 4, respectively, and 28 subjects in Cohort 6, will be dosed at least 3 days after the sentinel cohort.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the USA) prior to any study specific procedures.
* Male and/or female subjects aged 18 to 55 years (for Cohort 6 see below), inclusive, at the Screening Visit.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit/study site, must not be lactating and must be of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide starting from the time of IMP administration until 3 months after the final Follow-up Visit. It is strongly recommended for the female partner of a male subject to also use a highly effective method of contraception throughout this period.
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive, at the Screening Visit.
* Ability and willingness to adhere to the visit/protocol schedule and complete the Follow-up Period.

The subjects in Cohort 5 (subjects of Japanese descent) must fulfil the following additional criterion:

• Subjects must be of Japanese descent, defined as having 4 grandparents who are Japanese. This includes second and third generation subjects of Japanese descent whose parents or grandparents are living in a country other than Japan.

The subjects in Cohort 6 (subjects with CKD) must fulfil the following additional criteria:

* Male and/or female subjects aged 18 to 70 years, inclusive, at the Screening Visit.
* Have a BMI between 18 and 45 kg/m2 inclusive and weigh at least 50 kg and no more than 150 kg inclusive, at the Screening Visit.
* Subjects must have CKD, defined as:

  1. An estimated glomerular filtration rate (eGFR) 30 to 89 mL/min/1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, and
  2. Macroalbuminuria, defined as 300-3000 mg albumin/g creatinine based on the spot urine sample collected at the Screening Visit and the geometric mean of 3 sequential first morning void urine sample s at Visit 2 (Day 1).
* Stable BP meeting all of the following criteria:

  1. BP ≤ 150/100 mmHg at the Screening Visit and Visit 2 (Day -1).
  2. A stable dose of Angiotensin converting enzyme inhibitors (ACEi) or Angiotensin receptor blockers (ARB) for at least 4 weeks prior to the Screening Visit, per the local/site guidelines. Subjects who have been deemed unable to tolerate ACEi or ARB therapy due to allergy or complications may be enrolled. Dose adjustment of the next/previous titration dose within 2 weeks of the Screening Visit is acceptable.
  3. A stable dose of any other antihypertensive medication (including diuretic therapy) for at least 4 weeks prior to the Screening Visit.

Exclusion Criteria:

* History of any disease or condition that, in the opinion of the site PI and/or medical monitor, would place the subject at an unacceptable risk to participate in this study or interfere with evaluation of the investigational product or interpretation of subject safety or study results, including, but not limited to:

  1. History of any blood brain barrier (BBB) breakdown such as, but not limited to, recent traumatic brain/spinal injury, multiple sclerosis, active central nervous system vasculitis, recent stroke or cerebral hemorrhage, neurosurgery, meningoencephalitis, active or uncontrolled seizures, or lumbar puncture within the preceding 6 months.
  2. Prior malignancy other than non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy (response duration of > 5 years).
  3. Subjects with renal allografts.
* Proliferative retinopathy confirmed by retinal imaging at the Screening Visit
* History or presence of hematological, hepatic or renal disease (except Cohort 6) or any other condition known to interfere with administration, absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Any clinically relevant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening or Day -1 that, in the opinion of the site PI or medical monitor, may compromise the safety of the subject in the study, interfere with the evaluation of the IMP, or reduce the subjects' ability to participate in the study.

Note: Abnormal urinary findings will not exclude subjects in Cohort 6.

* Any laboratory values with the following deviations at screening or admission (for Cohort 6 see below):

  1. ALT > Upper limit of normal (ULN).
  2. AST > ULN.
  3. Total bilirubin (TBL) > ULN (unless due to Gilbert's syndrome).
  4. Creatinine > ULN.
  5. WBC count < lower limit of normal (LLN).
  6. Hb < LLN.
  7. Impaired renal function, defined as eGFR < 90 mL/min/1.73 m2 based on the CKD-EPI equation.
* Any positive result at the Screening Visit for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).
* Abnormal vital signs at Screening or Visit 2 (Day -1), after 10 minutes supine rest, defined as any of the following:

  1. SBP < 90 mmHg or ≥ 140 mmHg.
  2. DBP < 50 mmHg or ≥ 90 mmHg.
  3. HR < 45 or > 85 beats per minute (bpm).
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting 12-lead ECG as considered by the site PI that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy, at screening or admission.

  1. Prolonged QTcF > 450 ms.
  2. Family history of long QT syndrome.
  3. PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
  4. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
  5. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 120 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
* Known or suspected history of drug abuse as judged by the site PI.
* History of alcohol and/or substance abuse within the last 6 months or excessive intake of alcohol as judged by the site PI.
* Positive screen for drugs of abuse, including recreational marijuana, at the Screening Visit or upon admission to the Clinical Unit/study. Subjects who utilize benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the site PI or history of hypersensitivity to drugs with a similar chemical structure or class to MEDI8367.

  1. History of severe allergic reaction requiring hospitalization or,
  2. History of severe reaction to any medication including biologic agents or human gamma globulin therapy or,
  3. History of allergy or reaction to any component of the IMP formulation.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals with the 2 weeks or 5 half-lives prior to the first administration of IMP (Day 1) (whichever is longer). Further clarification regarding specific medications is provided below:

  1. Female subjects will be allowed to take hormone replacement therapy.
  2. Current or previous use of systemic corticosteroids within 60 days prior to Day 1 is prohibited
  3. Topical, intra-articular, nasal, inhaled, and ophthalmic corticosteroids are permitted.
  4. Antiplatelet therapy (i.e., aspirin, clopidogrel [Plavix], ticagrelor [Brilinta], or prasugrel), anticoagulation therapy (i.e., warfarin, factor Xa inhibitors, direct thrombin inhibitors, or heparin), and thrombolytic use, in the past month prior to Day 1 or planned use during the duration of the study, are prohibited.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to Day 1 (or > 1200 mL in the year prior to Day 1).
* Has received another new chemical or biologic entity (defined as a compound which has not been approved for marketing) within 4 months or 5 half-lives prior to the Screening Visit (whichever is longer), or planned participation in such a study prior to the end of the follow-up period.

Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.

* Scheduled surgery, including dental surgery, within 8 weeks of the scheduled completion date of the study.
* Involvement of any AstraZeneca, Clinical Unit, Contract Research Organization (CRO), or study site employee or their close relatives, regardless of the employee's role.
* Judgement by the site PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the site PI.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

The following exclusion criteria apply to subjects in Cohort 6 (subjects with CKD):

* Clinically significant late diabetic complications, including symptoms consistent with angina, congestive heart failure, and peripheral arterial disease (claudication), or other complications such as proliferative retinopathy, maculopathy, or gastroparesis.
* Chronic kidney disease due to abnormal anatomy of the urinary system or autosomal dominant polycystic kidney disease (ADPKD).
* Aggressive or serious neuropathies, in particular immune related demyelinating neuropathies such as Guillain-Barré, or one of its variants.
* Any laboratory values with the following deviations at screening or admission:

  1. ALT > 2 x ULN.
  2. AST > 2 x ULN.
  3. TBL > ULN (unless due to Gilbert's syndrome).
  4. Hb <100 g/L
  5. Glycated hemoglobin (HbA1C) > 10.5% measured at the Screening Visit.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals with the 2 weeks or 5 half-lives prior to the first administration of IMP (Day 1) (whichever is longer). Further clarification regarding specific medications is provided below:

  1. Subjects may take their usual prescribed medication, or any other medication taken on the advice of their physician with the exception of systemic corticosteroids. They should have been on a stable drug regimen with no changes in agents or doses for at least 4 weeks prior to participation in the study. Dose adjustment of the next/previous titration dose within 2 weeks of the Screening Visit is acceptable.
  2. Any serum creatinine-altering drugs within 1 month prior to the Screening Visit including but not limited to amphotericin, cimetidine, clofibrate, dronedarone, ketoconazole, probenecid, ranolazine, trimethoprim, aminoglycosides, or cephalosporins are prohibited.
  3. Use of insulin is prohibited.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to follow-up period (Day 90 ± 4 days)
  To assess AEs as a variable of safety and tolerability of SC of MEDI8367
Number of subjects with abnormal systolic blood pressure (SBP) | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess supine position SBP as a variable of safety and tolerability of MEDI8367
Number of patients with abnormal diastolic blood pressure (DBP) | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess supine position DBP as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal HR | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess change in supine position HR as a variable of safety and tolerability of MEDI8367
Number of subjects with respiratory rate | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess change in supine position respiratory rate as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal oral body temperature | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess change in oral body temperature as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal electrocardiogram (ECG) | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess electrical activity changes in ECG as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal physical examination | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess change in physical examination as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal structured neurological assessment | From screening (Day -28 ) up to follow-up period (Day 90 ± 4 days)
  To assess change in structured neurological assessment as safety and tolerability of MEDI8367. Any new or aggravated clinically relevant abnormal neurological examination finding compared to the baseline assessment will be reported as an AE
Number of subjets with abnormal retinal imaging | From screening (Day -28) up to follow-up period (Day 90 ± 4 days)
  To assess retinal imaging as a variable of safety and tolerability of MEDI8367. The presence of proliferative retinopathy or any other new retinal changes will be recorded. Any new or aggravated clinically relevant abnormal retinal imaging finding compared to the baseline assessment will be reported as an AE
Number of subjects with abnormal Hemoglobin (Hb) level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in Hb as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal red blood cells (RBC) count | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess RBC count as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal white blood cells (WBC) count | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess WBC count as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal differential WBC count | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess differential WBC count as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal hematocrit (HCT) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess HCT as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal mean corpuscular volume (MCV) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess MCV as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal mean corpuscular hemoglobin (MCH) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess MCH as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal reticulocytes absolute count | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess reticulocytes absolute count as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal mean corpuscular hemoglobin concentration (MCHC) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess MCHC as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal platelets count | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess platelets count as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal creatinine level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess creatinine level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal blood urea nitrogen level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess blood urea nitrogen level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urea level. | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses urea level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal bicarbonate level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses bicarbonate level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal creatine kinase (CK) level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses CK level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal follicle stimulating hormone (FSH)/luteinizing hormone (LH) level | From screening (Day -28) to treatment period (Day -1)
  To asses FSH/LH level for postmenopausal females as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal C-reactive protein (CRP) level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses CRP level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal cystatin C level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses cystatin C level in Cohort 6 only (subjects with CKD) as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal glucose (fasting) level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To asses glucose (fasting) level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal potassium level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess potassium level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal sodium level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess sodium level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal phosphate level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess phosphate level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal calcium level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess calcium level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal chloride level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess chloride level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal alkaline phosphatase (ALP) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess ALP level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal bilirubin level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess bilirubin level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal alanine aminotransferase (ALT) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess ALT as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal aspartate aminotransferase (AST) | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess AST as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal albumin level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess albumin level as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine protein level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine protein as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine glucose level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess changes in abnormal urine glucose as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine pH | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine pH as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine ketone level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine ketone as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine bilirubin level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine bilirubin as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine blood level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine blood as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine color. | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine color as a variable of safety and tolerability of MEDI8367 following SC administration of SAD.
Number of subjects with abnormal urine appearance. | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine apperance as a variable of safety and tolerability of MEDI8367 following SC administration of SAD.
Number of subjects with abnormal urine specific gravity level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine specific gravity as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine leukocyte esterase level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine leukocyte esterase as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine urobilinogen level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine urobilinogen as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine nitrite level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine nitrite as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine RBC level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine microscopy included RBC as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine WBC level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine microscopy included WBC as a variable of safety and tolerability of MEDI8367
Number of subjects with abnormal urine casts level | From screening (Day -28 to Day -2) through follow-up period (up to Day 90 ± 4 days)
  To assess change in urine microscopy casts as a variable of safety and tolerability of MEDI8367

SECONDARY OUTCOMES:
Plasma PK analysis: Maximum observed serum drug concentration (Cmax) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess Cmax of MEDI8367 following SC administration of SAD
Plasma PK analysis: Time to reach maximum observed concentration (tmax) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess tmax of MEDI8367 following SC administration of SAD
Plasma PK analysis: Terminal half-life (t½) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess t½ of MEDI8367 following SC administration of SAD
Plasma PK analysis: Area under the plasma concentration-time curve from zero to the last quantifiable concentration (AUClast) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess AUClast of MEDI8367 following SC administration of SAD
Plasma PK analysis: Area under plasma concentration-time curve from zero to infinity (AUCinf) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess AUCinf of MEDI8367 following SC administration of SAD
Plasma PK analysis: Apparent total body clearance of drug from serum after extravascular administration (CL/F) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess CL/F of MEDI8367 following SC administration of SAD
Plasma PK analysis: Volume of distribution (apparent) following extravascular administration (based on terminal phase; Vz/F) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess Vz/F of MEDI8367 following SC administration of SAD
Plasma PK analysis: Volume of distribution (apparent) at steady state following extravascular administration (Vss/F) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess Vss/F of MEDI8367 following SC administration of SAD
Plasma PK analysis: Area under plasma concentration-time curve from zero to the last quantifiable concentration divided by the dose administered (AUClast/D) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess AUClast/D of MEDI8367 following SC administration of SAD
Plasma PK analysis: Area under plasma concentration-time curve from zero to infinity divided by the dose administered (AUCinf/D) | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess AUCinf/D of MEDI8367 following SC administration of SAD
Plasma PK analysis: Maximum observed serum drug concentration divided by the dose administered (Cmax/D). | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess Cmax/D of MEDI8367 following SC administration of SAD.
Immunogenecity: ADA titer | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess ADA titer of MEDI8367 following SC administration of SAD
Immunogenecity: Anti-drug antibody (ADA) incidence. | From treatment period (Day 1) to follow-up period (up to Day 90 ± 4 days)
  To assess ADA incidence of MEDI8367 following SC administration of SAD.

CONTACTS AND LOCATIONS:
Overall Officials: Dr David Han, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home